CLINICAL TRIAL: NCT00585949
Title: The Effects of Age on Endothelial Progenitor Cell Mobilization in Humans
Brief Title: Age and Endothelial Progenitor Cell Mobilization
Acronym: AGE-PCI
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: American Federation for Aging Research (Other)
Responsible Party: Principal Investigator, Kreton Mavromatis, MD, FACC, Associate Professor, Emory University
Other Study IDs: IRB00045878
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon, Coronary; Cerebral Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Angiography: Patients undergoing coronary angiography without percutaneous coronary angioplasty
  Interventions: Procedure: Angiography
- Percutaneous Coronary Angioplasty: Patients with stable coronary artery disease undergoing angioplasty
  Interventions: Procedure: Percutaneous Coronary Angioplasty

INTERVENTIONS:
Procedure: Percutaneous Coronary Angioplasty — This is a procedure by which the blood vessels of the heart are imaged with an insertion of a catheter in the groin and blocked arteries are opened.
  Groups: Percutaneous Coronary Angioplasty
Procedure: Angiography — Angiography is an imaging technique to see coronary blood vessels.
  Groups: Angiography

SUMMARY:
It is hypothesized that aging is associated with reduced vascular injury-induced endothelial progenitor cell activity, resulting in impaired vascular repair and increased vascular disease. Patients with stable coronary artery disease will be enrolled in this observational study and will undergo either angiography alone or angiography and angioplasty. Participants will be followed for 5 years.

DETAILED DESCRIPTION:
Coronary artery disease is a leading cause of morbidity and mortality in our society. It is initiated by the dysfunction of the lining of coronary arteries. Such endothelial dysfunction permits vascular wall inflammation, smooth muscle cell proliferation, and thrombosis, which progresses to coronary artery stenosis and occlusion, and manifests as myocardial ischemia and infarction. Endothelial injury can be due to the damaging effects of various cardiovascular risk factors and it can also be induced by balloon injury associated with coronary angioplasty. Damaged endothelium can be repaired via endogenous mechanisms, such as by the migration and proliferation of neighboring uninjured mature endothelial cells, or by the mobilization and homing of bone-marrow-derived circulating endothelial progenitor cells (EPCs).

There are several repair mechanisms that are now thought to involve circulating endothelial progenitor cells that are mobilized from the bone marrow and home to sites of endothelial injury. The researchers of this study hypothesize that aging is associated with reduced vascular injury induced endothelial progenitor cell activity, resulting in impaired vascular repair and increased coronary heart disease events. Patients with stable coronary artery disease will be enrolled in this study. They will undergo either angiography alone or angiography and angioplasty. Venous blood will be collected immediately prior to the procedure and 20-24 hours after the procedure. The number of endothelial progenitor cells will be assessed based on their ability to form colonies and also to migrate under the influence of certain growth factors. These values will be compared between both samples. Study participants will also be contacted at 6 months, and 2 and 5 years after their participation in the study. The clinical outcomes of the participant's coronary artery disease will be correlated with the number of endothelial progenitor cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients having stable coronary artery disease and undergoing either angiography or angioplasty

Exclusion Criteria:

* Unstable coronary artery disease associated with either EKG changes or elevation of cardiac enzymes
* Coronary intervention in the past 3 months
* Renal insufficiency
* Malignancy within the past 5 years except non-melanomatous skin cancers
* Recent infection within the past 3 months requiring antibiotic treatment
* Recent surgery requiring anesthesia within the past 3 months
* Having inflammatory disease
* Chemotherapy, radiation therapy or bone marrow stimulants at any time in the past
* Menstruating women
* Recent changes in statin, angiotensin-converting enzyme (ACE) inhibitors, or angiotensin receptor blocker doses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stable coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10-09 (Actual); Study Completion 2008-10-09 (Actual)

PRIMARY OUTCOMES:
Change in endothelial progenitor cells colony forming units | 24 hours, 1 week, and 1 month after the procedure
  Activity of endothelial progenitor cells will be assessed in participants following their procedures.

SECONDARY OUTCOMES:
Change in clinical outcomes of coronary artery disease | Up to 5 years
  Participants will be contacted (or medical records will be examined) and asked if they have experienced cardiovascular disease outcomes such as myocardial infarction, stroke, hospitalization, coronary or peripheral revascularization, congestive heart failure exacerbation, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Kreton Mavromatis, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No